CLINICAL TRIAL: NCT07157891
Title: Investigating the Safety and Regenerative Potential of MSC-Derived Secretome Combined With PRGF in Knee Osteoarthritis
Acronym: PRGFSECKOA
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of the Punjab (Other)
Collaborators: Centre of Excellence in Molecular Biology (CEMB), University of the Punjab, Lahore. (Unknown)
Responsible Party: Principal Investigator, Noreen Latief, Assistant Professor, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSCSEC-OA-001
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis (OA); Knee Injury; Cartilage Degeneration
Keywords: Mesenchymal Stem Cell Secretome; Plasma Rich in Growth Factors (PRGF); Platelet-Rich Plasma (PRP); Knee Osteoarthritis; Intra-articular Injection; Cell-free Therapy; Regenerative Medicine
MeSH Terms: conditions — Osteoarthritis; Knee Injuries; Osteoarthritis, Knee | interventions — Culture Media, Conditioned

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC-Derived Secretome (Experimental): MSC-derived secretome will be administered as intra-articular injections under ultrasound guidance to the affected knee. Injection will be given twice, each after 6 months. Each injection will consist of 2 mL of concentrated MSC-derived secretome.
  Interventions: Biological: MSC-Derived Secretome
- MSC-Derived Secretome + Autologous PRGF (Experimental): MSC-derived secretome combined with autologous plasma-rich in growth factors plasma (PRGF) will be administered as intra-articular injections under ultrasound guidance to the affected knee. Injections will be given twice, each after 6 months. Each injection will consist of 2 mL of concentrated MSC-derived secretome and 1 mL of autologous PRGF, totaling 3 mL per dose.
  Interventions: Biological: MSC-Derived Secretome + Autologous PRGF

INTERVENTIONS:
Biological: MSC-Derived Secretome — The secretome will be collected from cultured MSCs under sterile, GMP-compliant conditions and concentrated to retain bioactive molecules. It will be injected into the affected knee under ultrasound guidance.
  Other Names: Conditioned Medium; MSC Secretome Therapy
  Arms: MSC-Derived Secretome
Biological: MSC-Derived Secretome + Autologous PRGF — MSC-derived secretome will be collected from mesenchymal stem cell cultures under sterile, GMP-compliant conditions. Autologous PRP will be prepared from the participant's own peripheral blood using a standardized single-spin centrifugation method and combined with 10% calcium chloride to activate growth factors. Both components will be mixed and administered into the affected joint under ultrasound guidance.
  Other Names: MSC-Secretome/PRGF Combined Therapy
  Arms: MSC-Derived Secretome + Autologous PRGF

SUMMARY:
This Phase I/II randomized clinical trial investigates the safety, feasibility, and early regenerative potential of intra-articular administration of mesenchymal stem cell (MSC)-derived secretome combined with Plasma Rich in Growth Factors (PRGF) in patients with knee osteoarthritis (KOA). The study aims to assess whether this cell-free, biologically enriched therapeutic combination can reduce pain, improve joint function, and promote cartilage repair.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic, degenerative joint disease characterized by progressive cartilage degradation, joint space narrowing, subchondral bone remodeling, inflammation, and pain that ultimately impair mobility and quality of life. Current treatment options, including analgesics, corticosteroids, and surgery, offer symptomatic relief but do not halt disease progression or restore joint tissue integrity.

Recent advancements in regenerative medicine have highlighted the therapeutic potential of mesenchymal stem cells (MSCs), particularly adipose-derived MSCs (AD-MSCs) and umbilical cord- derived MSCs (UC-MSCs), due to their robust paracrine activity. Rather than relying solely on cell engraftment, MSCs exert their therapeutic effects primarily through their secretome. These are complex mixtures of cytokines, growth factors, extracellular vesicles (EVs), and exosomes. This secretome can promote cartilage repair, reduce inflammation, and modulate immune responses, all without the risks associated with live cell transplantation.

This prospective, interventional study aims to evaluate the safety, tolerability, and early efficacy of intra-articular administration of MSC-derived secretome combined with Plasma Rich in Growth Factors (PRGF) in patients with mild to moderate symptomatic knee osteoarthritis (Kellgren-Lawrence grade II-III).The secretome will be collected from culture of human ADMSCs and UCMSCs grown in GMP-compliant labs, characterized for sterility, protein content, particle size, and bioactivity prior to administration.

Primary outcomes will include pain reduction assessment and any adverse events via Visual Analog Scale (VAS) and WOMAC index. If there will be adverse events, they will also be checked. Secondary outcomes will include functional improvement, cartilage regeneration (X-ray or MRI assessment), and changes in synovial inflammatory biomarkers (e.g., IL-1β, TNF-α, IL-6, MMP-13).

This study hypothesizes that the cell-free combination of MSC secretome and PRGF will offer regenerative benefits in knee OA, potentially improving joint function and structure while minimizing the risks associated with live cell therapies. Findings from this trial will inform the design of future large-scale studies and support the development of secretome-based regenerative therapies for osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Following is the inclusion criteria for the enrolment of patients affected with damaged cartilage in this study:

  * Diagnosed with primary OA in one or both knees based on American College of Rheumatology criteria
  * Grade I and II Arthritis
  * Joint pain ≥ 20mm measured by visual analogue scale
  * Age ranges from 30-55 years of age
  * BMI 27.12 ± 4.38
  * Patients with no previous surgical interventions to lower limb
  * Willing to participate in the study

Exclusion Criteria:

* • Secondary OA due to trauma, infection, rheumatoid arthritis, congenital disease or other inflammatory disorders of the knee

  * Diagnosed with a systemic autoimmune disorder, immunodeficiency or coagulation disorder
  * Had history of malignancy
  * History of allergy or allergic constitution
  * Pregnant or breastfeeding women.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-12-11 (Estimated); Study Completion 2028-12-11 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Pain (VAS Score) Change in WOMAC Score Adverse Events (Safety Monitoring) | From enrollment through the treatment period (Day 0 to Day 14); and at follow-up visits at 1 month, 3 months, 6 months, and 12 months post-treatment.
  Participants are evaluated for change in pain intensity using the Visual Analog Scale (VAS). Best outcome: pain score significantly reduced. If any Worst outcome: no change or increased pain.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) will be used to assess pain, stiffness, and physical function. Best outcome: improved total WOMAC score.
  Any local or systemic adverse events related to intra-articular administration of MSC secretome + PRP will be monitored and documented. Events will be categorized by type, severity, and relation to treatment.

OTHER OUTCOMES:
Change in Cartilage Thickness (MRI) Synovial Fluid Biomarkers Patient Global Assessment | From enrollment through the treatment period (Day 0 to Day 14); and at follow-up visits at 1 month, 3 months, 6 months, and 12 months post-treatment.
  Evaluation of articular cartilage thickness, signal intensity, and subchondral bone integrity using MRI. Best outcome: increased or preserved cartilage thickness, reduced signal abnormalities.
  Quantification of inflammatory biomarkers (e.g., IL-1β, TNF-α, MMP-13) in synovial fluid to assess joint inflammation. Best outcome: significant reduction in pro-inflammatory marker levels post-treatment.
  Self-reported patient evaluation of symptom relief and joint mobility using a standardized global assessment scale. Best outcome: improved self-perceived joint health.

IPD SHARING:
Plan to Share IPD: Undecided